CLINICAL TRIAL: NCT04140747
Title: Transfer of Strictly Anaerobe Microbes From Mother to Child - a Pilot Study
Brief Title: Transfer of Strictly Anaerobe Microbes From Mother to Child
Acronym: TRAMIC
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 28-524 ex 15/16
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — from non-pregnant and pregnant women: serum, urine, oral swabs, vaginal swabs, stool
  from pregnant women undergoing C-section: amniotic fluid
  from newborn babies: cord blood, oral swabs, meconium, stool sample of day 1-3
  colostrum and breast milk samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-pregnant women: Samples will be collected from 30 healthy, non-pregnant women in the reproductive age: blood, urine, stool, saliva, oral swabs, vaginal swabs
- pregnant women delivering vaginally: From 30 healthy, pregnant women giving vaginal birth, samples will be collected shortly before, during and after birth from maternal and newborn sites:
  maternal blood, urine, stool, saliva, oral swabs, vaginal swabs; cord blood, colostrum, meconium, infant oral swabs
- pregnant women undergoing C-section: From 30 healthy, pregnant women giving vaginal birth, samples will be collected shortly before, during and after birth from maternal and newborn sites:
  maternal blood, urine, stool, saliva, oral swabs, vaginal swabs; amniotic fluid, cord blood, colostrum, meconium, infant oral swabs

SUMMARY:
This study aims to investigate the changes in the microbiota at different body sites in late pregnancy, in comparison with non-pregnant women, with particular emphasis on archaea, and to identify possible maternal-to-child transfer routes for acquisition of strictly anaerobic microorganisms by analyzing the gut microbiota of new born infants (delivered vaginally or by C-section).

DETAILED DESCRIPTION:
The investigators hypothesize that changes occur in the microbial community during pregnancy in different body sites (vagina, oral etc.) and that the main source of these microorganisms is the mother for vaginally born infants, while C-section born infants acquire most of the anaerobic microbial communities from other sources rather than mother's vaginal and gut microbiota, such as the environment.

Specific Research Objectives will be:

1. To investigate diversity of archaea in the vagina of healthy women in the context with community state types (CSTs), and compare vaginal microbiome in pregnant with non-pregnant healthy women.
2. To identify the presence of archaea in different body sites (oral, gut) or body fluids (amniotic fluid, urine, human milk) within the perinatal microbial communities.
3. To investigate the presence of archaea in the infant's first-days-of-life intestinal community, and to identify the sources of these microorganisms by using source tracking approach.
4. To investigate Human Milk Oligosaccharides (HMOs) in maternal (serum, saliva, urine, breast milk) or intrauterine sources (amniotic fluid) as potential modifiers of the microbial communities in these sites.
5. To analyze associations of maternal/ intrauterine HMOs with infant HMOs and microbiota (meconium and infant stool) in order to investigate vertical transmission of microbiota to the infant.

ELIGIBILITY:
Inclusion Criteria:

* healthy women
* pregnant women: delivery at term (gestational age 37-42); contractions or rupture of membrane no longer than 12h before admission to hospital

Exclusion Criteria:

* bacterial/ fungal infections
* use of antibiotics/ probiotics in past 3 months
* fetal anomalies
* multiple pregnancies
* diabetes type 1, 2, gestational diabetes
* hypertension, preeclampsia/HELLP
* HIV ( human immunodeficiency virus), HCV (Hepatitis C)
* drug abuse, smoking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy non-pregnant women and women with an ongoing healthy pregnancy. 3 groups will be formed: non-pregnant women (n=30), women delivering vaginally (n=30) and women undergoing C-section (n=30).
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
maternal microbiome | 2020-2023
  difference between non-pregnant and pregnant women
fetal/neonatal microbiome | 2020-2023
  difference between vaginal and C-section born infants

SECONDARY OUTCOMES:
Human milk oligosaccharides | 2020-2023
  associations of HMOs with maternal/infant microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Jantscher-Krenn, PhD, Principal Investigator — Medical University of Graz; Christine Moissl-Eichinger, PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria